CLINICAL TRIAL: NCT05777694
Title: Investigation of the Effect of Needle Thickness on Postdural Puncture Headache: a Prospective Randomized Study
Brief Title: Postdural Punction Headache After Ceserian Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-297
Record Dates: First submitted 2023-02-24; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Postdural Puncture Headache; Regional Anesthesia Morbidity; Pregnancy Related
Keywords: cesarean section; obstetric anesthesia; spinal anaesthesia; postdural punction headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Intervention Model Description: pospective randomize study
Masking Description: The prospective randomized study was randomized into 3 groups:
  Group 1: Patients who underwent cesarean section under spinal anesthesia with 25 gauge spinal needle ( Pencan® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany) Group 2: Patients who underwent cesarean section under spinal anesthesia with 26 gauge spinal needle ( Atraucan® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany) Group 3: Patients who underwent cesarean section operation under spinal anesthesia with 27 gauge spinal needle ( Pencan ® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: 25 gauge spinal needle (Active Comparator): Group 1: Patients who underwent cesarean section under spinal anesthesia with 25 gauge spinal needle ( Pencan® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany)
  Interventions: Procedure: Patients who underwent cesarean section under spinal anesthesia with 25 gauge spinal needle; Procedure: Patients who underwent cesarean section under spinal anesthesia with 26 gauge spinal needle; Procedure: Patients who underwent cesarean section operation under spinal anesthesia with 27 gauge spinal needle
- Group 2: 26 gauge spinal needle (Active Comparator): Group 2: Patients who underwent cesarean section under spinal anesthesia with 26 gauge spinal needle ( Atraucan® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany)
  Interventions: Procedure: Patients who underwent cesarean section under spinal anesthesia with 25 gauge spinal needle; Procedure: Patients who underwent cesarean section under spinal anesthesia with 26 gauge spinal needle; Procedure: Patients who underwent cesarean section operation under spinal anesthesia with 27 gauge spinal needle
- Group 3: 27 gauge spina needle (Active Comparator): Group 3: Patients who underwent cesarean section operation under spinal anesthesia with 27 gauge spinal needle ( Pencan ® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany)
  Interventions: Procedure: Patients who underwent cesarean section under spinal anesthesia with 25 gauge spinal needle; Procedure: Patients who underwent cesarean section under spinal anesthesia with 26 gauge spinal needle; Procedure: Patients who underwent cesarean section operation under spinal anesthesia with 27 gauge spinal needle

INTERVENTIONS:
Procedure: Patients who underwent cesarean section under spinal anesthesia with 25 gauge spinal needle — the investigators performed spinal anesthesia with 25 gauge pencil point spinal needle to that patient group for prevent postdural puncture headache
Procedure: Patients who underwent cesarean section under spinal anesthesia with 26 gauge spinal needle — the investigators performed spinal anesthesia with 26 gauge pencil point spinal needle to that patient group for prevent postdural puncture headache
Procedure: Patients who underwent cesarean section operation under spinal anesthesia with 27 gauge spinal needle — the investigators performed spinal anesthesia with 27 gauge pencil point spinal needle to that patient group for prevent postdural puncture headache

SUMMARY:
The aim of this study is to compare the effect of spinal needle type on postdural puncture headache in patients who will undergo cesarean section.

The main question[s] it aims to answer are:

[Does spinal needle thickness affect postdural puncture headache?]

[What is the response of patients who develop postdural puncture headache to treatment?] In cases accepting cesarean section operation under spinal anesthesia, different tables were used with spinal needles, and it will be questioned whether headache will develop in the first 15 days postoperatively. Postdural puncture headache after surgery will be described.

DETAILED DESCRIPTION:
Our study was designed as a prospective randomized study. Patients aged 20-50 years who accepted cesarean section under elective spinal anesthesia were included in the study. randomized into 3 groups with 250 patients in each group:

Group 1: Patients who underwent cesarean section under spinal anesthesia with 25 gauge spinal needle ( Pencan® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany) Group 2: Patients who underwent cesarean section under spinal anesthesia with 26 gauge spinal needle ( Atraucan® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany) Group 3: Patients who underwent cesarean section operation under spinal anesthesia with 27 gauge spinal needle ( Pencan ® 0.42 × 88 mm- G27 × 3½, B. Braun, Melsungen, Germany) Postdural puncture headache (PDPH) was evaluated by visiting patients who were discharged to the service after spinal anesthesia in the hospital for 24 hours, and by calling them within 15 days after discharge. Conservative and medical treatment was recommended for patients who developed PDPH, and the response of the patients to treatment was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who accept spinal anesthesia and have no contraindications for spinal anesthesia Ages of 20-50 years ASA II-III

Exclusion Criteria:

* Pregnant women who do not accept spinal anesthesia and who are contraindicated for spinal anesthesia Morbid obesity(BMI>40) Coagulopaty ASA 4 Clinically known local anesthetic allergy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 750 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
PDPH and spinal needle | postoperatively 15 days. The hospital was visited on the first day and information was obtained by calling in the following days. Patients with PDPH were evaluated as mild (1-3), moderate (4-7), severe (8-10) according to the Lybecker classification.
  The primary aim of this study is to investigate the effect of needle type used on postdural puncture headache.

SECONDARY OUTCOMES:
Treatment response of patients with PDPH | postoperatively 15 days, The hospital was visited on the first day and information was obtained by calling in the following days. Oral drugs used in the treatment and recommendations were noted.
  Response rate of patients with PDPH to conservative and medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akyol, M.D, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient data will be kept confidential.

REFERENCES:
- [Result] Chekol B, Yetneberk T, Teshome D. Prevalence and associated factors of post dural puncture headache among parturients who underwent cesarean section with spinal anesthesia: A systemic review and meta-analysis, 2021. Ann Med Surg (Lond). 2021 Jun 2;66:102456. doi: 10.1016/j.amsu.2021.102456. eCollection 2021 Jun. PMID 34141426
- [Result] Lee SI, Sandhu S, Djulbegovic B, Mhaskar RS. Impact of spinal needle type on postdural puncture headache among women undergoing Cesarean section surgery under spinal anesthesia: A meta-analysis. J Evid Based Med. 2018 Aug;11(3):136-144. doi: 10.1111/jebm.12311. Epub 2018 Aug 1. PMID 30070060
- [Result] Mowafy SMS, Ellatif SEA. Effectiveness of nebulized dexmedetomidine for treatment of post-dural puncture headache in parturients undergoing elective cesarean section under spinal anesthesia: a randomized controlled study. J Anesth. 2021 Aug;35(4):515-524. doi: 10.1007/s00540-021-02944-6. Epub 2021 May 16. PMID 33993346